CLINICAL TRIAL: NCT00720889
Title: Sleep, Energy Metabolism and Diabetes Risk.
Brief Title: Glucose Metabolism and Sleep in People With Family History of Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16079A-S2; R01HL089637 (NIH)
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sleep; Insulin Resistance; Type 2 Diabetes
Keywords: short sleep duration; glucose clamp technique; insulin secretion; insulin action; lipid turnover; free fatty acids
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Reduced sleep: Habitual sleep duration of less than 6 hours per night on most days of the week and total sleep of less than 43 hours per week.
- Reference sleep: Habitual sleep duration between 7 and 8.5 hours per night on most days of the week and total sleep of at least 53 hours per week.

SUMMARY:
The use of sugar and starch-like foods for energy (carbohydrate metabolism) changes when people sleep. However, it is still not known if differences in the amount of nighttime sleep have an effect on the carbohydrate metabolism of people who have a relative with type 2 diabetes (parent, sibling, or grandparent). This study is being done to test the hypothesis that individual differences in habitual sleep duration may be related to differences in the carbohydrate metabolism of people who have a history of type 2 diabetes in their family.

DETAILED DESCRIPTION:
On two consecutive inpatient days, the participants in this study will undergo two different tests. The first test will determine how much insulin can their body produce in response to an intravenous glucose infusion over a period of several hours. The second test will determine how effective is the action of the sugar-processing hormone, insulin, in their body when it is infused intravenously together with glucose over a period of several hours.

ELIGIBILITY:
Inclusion Criteria:

* regular sleep habits
* BMI 20 to 27 kg/m2
* at least one parent, sibling or grandparent with type 2 diabetes
* no regular exercise habits

Exclusion Criteria:

* active smoker
* night or shift work
* have highly variable sleep habits
* have a hormonal disorder
* have a sleep disorder
* have an active medical problem
* women only: use of birth control pills
* women only: irregular menstrual periods or pregnancy
* use of medications/compounds that can disrupt sleep

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy non-obese community-living men and women with a parent, sibling or grandparent who has type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total body insulin sensitivity | at the end of a 4-hour hyperinsulinemic clamp

SECONDARY OUTCOMES:
First and second phase insulin secretion | during a 3-hour hyperglycemic clamp
Endogenous glucose production | before and during a 4-hour hyperinsulinemic clamp
Glycerol turnover and free fatty acid concentration | before and during a 4-hour hyperinsulinemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Plamen D Penev, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States